CLINICAL TRIAL: NCT06704282
Title: Effects of VR-Based Mindfulness Observational Meditation for Stress Reduction in Adults : Randomized Controlled Trial
Brief Title: Assessing the Impact of VR-Based Observational Mindfulness Meditation on Stress Reduction in Adults
Acronym: VR-MOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, JiHeun Hong, Visiting Scholar, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00025978
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Stress; Anxiety; Depression
Keywords: Mindfulness; Virtual Reality; Meditation; Observe Activity
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the experimental group, receiving mindfulness-based VR observational meditation, or the control group, undergoing standard relaxation techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Meditation Group (Experimental): Participants in this arm will undergo a 15-minute VR-based mindfulness observational meditation session guided by a virtual coach. The intervention focuses on promoting mindfulness and reducing stress through structured guidance in a controlled virtual environment.
  Interventions: Behavioral: VR Mindfulness Meditation Program

INTERVENTIONS:
Behavioral: VR Mindfulness Meditation Program — A 15-minute guided mindfulness meditation session conducted in a virtual reality environment to enhance stress reduction and mindfulness.

SUMMARY:
This study investigates the impact of a mindfulness-based intervention using virtual reality (VR) and artificial intelligence (AI) coaching on stress reduction. Participants will engage in VR-based observation mindfulness activities guided by an AI coach. The study aims to evaluate the effectiveness of this intervention compared to a standard relaxation process by measuring self-reported stress levels, physiological biomarkers (e.g., heart rate), and participant satisfaction. The research could inform the development of future digital mental health interventions.

DETAILED DESCRIPTION:
This study employs a randomized controlled design to assess the effectiveness of a VR-based mindfulness intervention for stress reduction. Participants are randomly assigned to either the experimental group, which undergoes VR-based observation mindfulness activities guided by an AI coach, or the control group, which experiences standard relaxation exercises. Pre-intervention data, including self-reported stress levels (measured via PSS-10, DASS-21, and STAI) and baseline heart rate, are collected. Following the intervention, participants complete post-intervention measurements to evaluate changes in stress levels, physiological responses, and satisfaction with the VR program.

The experimental group participates in mindfulness activities designed to enhance attention to detail and present-moment awareness through object observation within the VR environment. The AI coach facilitates the session by prompting reflective and observational questions, fostering deeper engagement. The control group undergoes relaxation exercises with no active mindfulness engagement. All procedures are conducted in a controlled laboratory setting, ensuring consistency and minimizing external variables.

The study collects objective (heart rate and heart rate variability) and subjective (self-reported stress and satisfaction) data to evaluate the intervention's efficacy. The findings aim to provide insights into the feasibility and benefits of integrating VR and AI technologies in stress reduction interventions. The results will also contribute to the development of more engaging and accessible digital mindfulness practices for diverse populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.

Exclusion Criteria:

* Those with visual or hearing impairments that prevent interaction with VR content.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-23 (Estimated)

PRIMARY OUTCOMES:
Reduction in Perceived Stress Levels | Immediately post-intervention (Day 1, 15 minutes after the session ends).
  Changes in perceived stress levels measured using the Perceived Stress Scale (PSS-10) to assess the effectiveness of the VR-based mindfulness observational meditation intervention.
Changes in Emotional State | Immediately post-intervention (Day 1, 15 minutes after the session ends).
  Emotional state assessed using the Depression Anxiety Stress Scales (DASS-21) and the State-Trait Anxiety Inventory (STAI). These indicators will be evaluated pre- and post-intervention to measure reductions in anxiety and overall emotional improvement.
Participant Satisfaction with Intervention | Immediately post-intervention (Day 1).
  Participant satisfaction assessed via a structured satisfaction survey post-intervention, including feedback on usability, perceived effectiveness, and comfort with the VR program.
Physiological Stress Response | Baseline (before intervention) and immediately post-intervention (Day 1).
  Heart rate measured pre- and post-intervention using a heart rate monitor to assess changes in physiological stress levels as a biomarker.
Changes in Emotional State Using STAI | Baseline (prior to intervention) and immediately post-intervention (Day 1, 15 minutes after the session ends).
  Anxiety levels will be assessed using the State-Trait Anxiety Inventory (STAI), which measures both state and trait anxiety components. The STAI-S (State Anxiety) evaluates participants' current feelings, while the STAI-T (Trait Anxiety) measures participants' general tendencies toward anxiety. Measurements will be taken pre- and post-intervention to evaluate reductions in anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Univercity, Erie, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be made available upon request. All shared data will be fully anonymized to protect participant confidentiality and privacy. Researchers can request access by contacting the primary investigator at the provided email address. Access will be granted for non-commercial research purposes only, subject to review and approval by the study team.

REFERENCES:
- [Derived] Hong J, Shelton CR, Oh H. Randomised controlled trial of VR-based observation meditation with AI coaching ('Otti') for stress reduction in university students in the United States: study protocol. BMJ Open. 2025 Oct 23;15(10):e097236. doi: 10.1136/bmjopen-2024-097236. PMID 41130677